CLINICAL TRIAL: NCT00825695
Title: Flavanol-Rich Cocoa, Vascular Responses and Mechanisms
Brief Title: Flavanol-Rich Cocoa and Cerebral Blood Flow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: MasterFoods (Industry)
Responsible Party: Principal Investigator, Naomi DL Fisher, MD, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: P-001936; 1R01HL089570 (NIH)
Record Dates: First submitted 2009-01-20; First posted 2009-01-21 (Estimated); Last update posted 2014-04-30 (Estimated); Status verified 2014-04

CONDITIONS: Hypertension; Diabetes
MeSH Terms: conditions — Hypertension; Diabetes Mellitus | interventions — Chocolate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- flavanol-rich cocoa (Active Comparator)
  Interventions: Dietary Supplement: cocoa
- flavanol-poor cocoa (Placebo Comparator)
  Interventions: Dietary Supplement: cocoa

INTERVENTIONS:
Dietary Supplement: cocoa — two servings of cocoa daily for one month
  Other Names: Cocoa Pro

SUMMARY:
The purpose of the study is to learn whether or not cocoa has a beneficial effect on blood flow to the brain in older subjects with diabetes mellitus or hypertension (high blood pressure). We hypothesize that cocoa, which contains flavanols (a type of polyphenol), may help to promote blood flow to the brain in older people with diabetes or hypertension.

ELIGIBILITY:
Inclusion Criteria:

* diabetes and/or hypertension

Exclusion Criteria:

* alzheimers disease, dementia, stroke, recent angina or heart attack

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-01; Primary Completion 2012-03 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
functional transcranial doppler measures | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Naomi D. Fisher, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States